CLINICAL TRIAL: NCT03087266
Title: Acute-phase Response Following Full-mouth Versus Quadrant Non-surgical Periodontal Treatment in Diabetes-affected Subjects: A Randomized Clinical Trial
Brief Title: Acute-phase Response & Periodontal Treatment in Diabetes Affected Patients
Acronym: PERIO-DIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Professor of Periodontology, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3399/11_A
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Periodontitis; Diabetes
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: single-centre randomized controlled clinical trial with a 3- month follow-up
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full- Mouth Scaling and Root Planing (Experimental): FM-SRP Non-surgical periodontal treatment will be performed in all dentition within 24 hours.
  Interventions: Procedure: FM-SRP
- Quadrant Scaling and Root Planing (Active Comparator): Q-SRP Non-surgical periodontal treatment will be performed in all dentition subdivided in four appointments. Each appointment will be performed with one week interval. In each appointment only a "quadrant" of the dentition will be instrumented.
  Interventions: Procedure: Q-SRP

INTERVENTIONS:
Procedure: FM-SRP — Non surgical periodontal treatment performed in all dentition within 1-2 appointments in a 24 hour time frame.
  Arms: Full- Mouth Scaling and Root Planing
Procedure: Q-SRP — Non surgical periodontal treatment performed in 4 sessions comprising of a quadrant (1/4) of the dentition each. Performed in 3 weeks time frame.
  Arms: Quadrant Scaling and Root Planing

SUMMARY:
Thirty-eight periodontitis- and diabetes-affected subjects will be randomly allocated to non surgical periodontal treatment with either Full-Mouth Approach (FM-SRP) or Quadrant approach (Q-SRP).

Patients will be seen one day and three months (study completion) after treatment. The 24 hours appointment will be occurring after the entire completion of the FM-SRP or the first quadrant of the Q-SRP. In the latter group other sessions of treatment will be performed within the following 3 weeks.

At baseline, 24 hours and three months, anthropometric, inflammatory and endothelial parameters will be collected. Periodontal parameters will be checked at baseline and at three months.

Main outcome of the study is the level of C-reactive protein 24 hours after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Periodontal disease
* 20% of periodontal pockets of the entire dentition
* 20% bleeding on probing of the entire dentition
* documented radiographic bone loss
* Diagnosis of Diabetes Type 2 as measured through international standards

Exclusion Criteria:

* age younger than 18 years and older than 80 years
* pregnant or lactating females
* females using contraceptive methods
* need of antibiotic coverage for periodontal treatment
* previous periodontal treatment in the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Levels C-Reactive Protein | Baseline, 24 hours and 3 months after treatment
  Changes in C reactive protein (CRP). Unit of measure: mg/L

SECONDARY OUTCOMES:
Full Mouth Plaque Score (FMPS) | Baseline and 3 months after treatment
  Changes in FMPS. Unit of Measure: %
Full Mouth Bleeding Score (FMBS) | Baseline and 3 months after treatment
  Changes in FMBS. Unit of Measure: %
Pocket probing depth (PPD) | Baseline and 3 months after treatment
  Changes in PPD. Unit of measure: mm
Clinical attachment level (CAL) | Baseline and 3 months after treatment
  Changes in CAL. Unit of measure: mm
Recession of the gingival margin (REC) | Baseline and 3 months after treatment
  Changes in REC. Unit of measure: mm
Triglycerides | Baseline, 24 hours and 3 months after treatment
  Changes in triglycerides. Unit of measure: mmol/L
Low-density lipoprotein (LDL) | Baseline, 24 hours and 3 months after treatment
  Changes in LDL. Unit of measure: mmol/L
High-density lipoprotein (HDL) | Baseline, 24 hours and 3 months after treatment
  Changes in HDL. Unit of measure: mmol/L
Cholesterol | Baseline, 24 hours and 3 months after treatment
  Changes in total cholesterol, Unit of measure: mmol/L
Glycemia | Baseline, 24 hours and 3 months after treatment
  Changes in blood glucose level. Unit of measure: mg/dl
Glycated Haemoglobin | Baseline, 24 hours and 3 months after treatment
  Changes in Glycated haemoglobin. Unit of measure: mmol/mol
Insulin | Baseline, 24 hours and 3 months after treatment
  Changes in Insulin level
Systolic Blood Pressure (SBP) | Baseline, 24 hours and 3 months after treatment
  Changes in SBP Unit of measure: mmHg
Diastolic Blood Pressure (DBP) | Baseline, 24 hours and 3 months after treatment
  Changes in DBP. Unit of measure: mmHg
Endothelial Function | Baseline, 24 hours and 3 months after treatment
  Measures of endothelial function taken through Flow-Mediated dilation. Unit of Measure: %

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Graziani, DDS, MClinDent, PhD, Principal Investigator — University of Pisa
Locations (1):
- University Hospital of Pisa, Pisa, Italy

REFERENCES:
- [Derived] Graziani F, Gennai S, Marruganti C, Peric M, Ghiadoni L, Marhl U, Petrini M. Acute-phase response following one-stage full-mouth versus quadrant non-surgical periodontal treatment in subjects with comorbid type 2 diabetes: A randomized clinical trial. J Clin Periodontol. 2023 Apr;50(4):487-499. doi: 10.1111/jcpe.13760. Epub 2023 Jan 22. PMID 36517997